CLINICAL TRIAL: NCT07379554
Title: Personalized Immunological Score for the Prediction of Severe Infectious Events in Immunocompromised Patients and Tailored Management (PERISCOPE)
Acronym: PERISCOPE
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Irene Cassaniti, PhD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: PERISCOPE
Record Dates: First submitted 2025-12-05; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-08

CONDITIONS: Immunocompromised Patients; Transplant Patients; Infections
Keywords: Immunological score; severe infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immunocompromised patients: We plan to prospectively enroll 150 immunocompromised patients during the first year of the study, including:
  * adult hematopoietic stem cell transplant recipients (a-HSCTR)
  * pediatric hematopoietic stem cell transplant recipients (p-HSCTR)
  * solid organ transplant recipients (SOTR), including kidney, heart and lung transplanted patients.

SUMMARY:
Transplants have improved clinical conditions for many patients with haematological diseases and end-stage organ diseases. However, immunosuppressive therapies that are necessary for avoiding organ rejection have a crucial impact in the occurrence of opportunistic infections. Despite the development of effective antimicrobial agents, infectious diseases are still related to mortality and morbidity in immunocompromised patients. Immune function assays can be adopted for monitoring T-cell function and eventually modify immunosuppression. Given the inverse relationship between cellular immune reconstitution and risk of infection, many transplant centers prospectively monitor immune recovery post-transplant. Some basic methods are useful, including white blood cells and T-lymphocyte subsets count. Given the complexity of immune responses required to resolve infections, functional assays are necessary and the only available FDA-approved one is Cyclex-Immuknow. Viral infections are common in patients with T-cell deficiencies and are of particular concern in those receiving high dose steroids. Opportunistic infections are common during the period of highest immunosuppression while community acquired infections, including fungal and respiratory viruses infections, have to be considered in the long-term period. Reduced CD4+ and CD8+ T-lymphocyte counts correlate with risk of opportunistic infection, including human cytomegalovirus (HCMV). Moreover, a decrease in human Rhinovirus (HRV) load in pediatric hematopoietic stem cell transplant recipients (HSCTRs) was associated with a significant increase in T-CD4+, T-CD8+ and NK lymphocytes, suggesting that cellular immunity have a crucial role in viral clearance and infectious control. A recent study showed that poor NK-cell cytotoxic activity is associated with increased risk for severe infections in kidney-graft recipients, suggesting that assessment of NK-cell function may be used as a predictor of infection in immunocompromised patients. Moreover, it has been recently reported that NKG2C genotype influences receptor function and NKG2C+ NK cell number in HCMV seropositive subjects. In detail, NKG2C genotype is significantly associated with HCMV viremia frequency and related disease after lung transplant and with symptomatic CMV infection after kidney transplant. Beside the use of non-specific immunological markers, the lack of standardized quantitative measures of protective immune functions specific for different opportunistic pathogens represents a challenge for clinicians. Overall, a comprehensive approach based on the use of combined non-specific and pathogen-specific immune assays may help in the definition of a composite immune risk profile of immunocompromised patients. The ultimate goal of this research is the definition of algorithms of infectious risk in immunocompromised patients, leading to a more adherent administration of immunosuppressive and antimicrobial therapies as well as to a personalized strategy of patients' management. Moreover, the design of new immunological assays that can be standardized and used in the clinical practice will be obtained.

Currently, even if an immunological monitoring of immunocompromised patients is recommended, no standardized assays and protocols are available, especially for the use of antigen-specific or functional assays. The introduction of diagnostics algorithms will be useful for the stratification of patients at high risk of infections that will be monitored more frequently in order to prevent severe infections. Similarly, the administration of immunosuppressive drugs or ad hoc therapies might be tailored according to the risk of infections or complications. Objective is to identify a composite immune score measured either before or one month after transplant/chemotherapy able to define the risk for clinically significant infections (e.g. infections requiring antimicrobial therapy or hospitalization) during the following three months.

Primary endpoint:

To identify a composite immune score measured either before or one month after transplant/chemotherapy able to define the risk for clinically significant infections (e.g. infections requiring antimicrobial therapy or hospitalization) during the following three months.

Secondary endpoints:

* To evaluate the prognostic effect of the immunological score measured before or at first month after transplant/chemotherapy on the risk of severe infection during the following 6-12 months
* To compare the role of the composite immunological score with specific assays against each pathogen.
* To develop simple and rapid assays using whole blood to evaluate specific pathogen responses

ELIGIBILITY:
Inclusion Criteria:

adult hematopoietic stem cell transplant recipients (a-HSCTR)

* pediatric hematopoietic stem cell transplant recipients (p-HSCTR)
* solid organ transplant recipients (SOTR), including kidney, heart and lung transplanted patients.

Written informed consent

Exclusion Criteria:

* no written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adult hematopoietic stem cell transplant recipients (a-HSCTR)
  * pediatric hematopoietic stem cell transplant recipients (p-HSCTR)
  * solid organ transplant recipients (SOTR), including kidney, heart and lung transplanted patients.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Immunological score for predicting severe infections | From enrolment to three months of follow up
  A composite immune score including overall number of T cells (CD3+CD4+, CD3+CD8+, CD3-CD56+NK cells, CD19+ B cells), Herpesviruses-specific T-cell response (e.g CMV, EBV, HSV1 and 2, VZV) measured before or one month after transplant/chemotherapy will be compared in patients with and without clinically significant infections (e.g. infections requiring antimicrobial therapy or hospitalization) registered during the following three months.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy